CLINICAL TRIAL: NCT07127458
Title: Prevalence of Anxiety and Depression in Adolescents With Polycystic Ovary Syndrome
Brief Title: Anxiety and Depression in Adolescent PCOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Sabahattin Anıl Arı, Associate Professor, Ege University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-PCOS-1
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-08

CONDITIONS: PCOS (Polycystic Ovary Syndrome)
Keywords: Polycystic Ovary Syndrome (PCOS); Adolescents; Anxiety and Depression
MeSH Terms: conditions — Polycystic Ovary Syndrome; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adolescents with Polycystic Ovary Syndrome (Experimental): Adolescent patients with PCOS will be identified, and the prevalence of anxiety and depression will be assessed. Oral contraceptive therapy will be initiated, and patients will be re-evaluated after 6 months.
  Interventions: Drug: Adolescent PCOS group receiving oral contraceptives

INTERVENTIONS:
Drug: Adolescent PCOS group receiving oral contraceptives — Participants diagnosed with polycystic ovary syndrome (PCOS) during adolescence will receive a combined oral contraceptive (ethinylestradiol 30 µg + drospirenone 3 mg) once daily for six consecutive months. The intervention aims to regulate menstrual cycles, reduce hyperandrogenic symptoms, and evaluate changes in anxiety and depression scores over time.

SUMMARY:
Polycystic ovary syndrome (PCOS) is a prevalent endocrine disorder in adolescent females, often accompanied by psychological symptoms such as anxiety and depression. These conditions are frequently underdiagnosed and untreated. This study aims to determine the prevalence of anxiety and depression in adolescents with PCOS and to assess changes following oral contraceptive use.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a common endocrine disorder in women of reproductive age, characterized by heterogeneous complications. It is increasingly prevalent among adolescent females today. Women with PCOS may experience infrequent or prolonged menstrual periods, excessive hair growth, acne, and obesity. The rising prevalence of PCOS in the general population affects approximately 5-10% of women of reproductive age worldwide (1). A significant proportion of women with PCOS-particularly adolescent girls-experience major depressive disorder. Although the exact cause of PCOS remains unknown, early diagnosis and treatment, along with weight loss, can reduce the risk of long-term complications. Depression and anxiety are common in women with PCOS; however, their frequency has often been overlooked, leaving many cases untreated (2). In addition to physical symptoms, various mental health problems are also associated with PCOS (3). The diagnosis of PCOS is established when at least two of the following criteria are present: amenorrhea/oligomenorrhea, hyperandrogenism (clinical or biochemical), and a polycystic ovarian appearance on ultrasound (4). Psychosocial problems are particularly common among obese adolescents and those with excessive hair growth.

The rationale of this study is to investigate the prevalence of this often-overlooked comorbidity and to evaluate changes following OCS (oral contraceptive) use.

ELIGIBILITY:
Inclusion Criteria:

* Age between 15 and 19 years
* Diagnosis of adolescent polycystic ovary syndrome (PCOS)

Exclusion Criteria:

* Severe reading or comprehension difficulties
* Severe hearing impairment
* Current use of hormone therapy
* Presence of a virilizing tumor
* Major psychiatric disorders such as schizophrenia, bipolar disorder, or dissociative disorder

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 42 (Estimated)
Dates: Start 2025-08-17 (Actual); Primary Completion 2026-03-17 (Estimated); Study Completion 2026-03-17 (Estimated)

PRIMARY OUTCOMES:
Change in Beck Depression Inventory | 6 Months
  Change in Beck Depression Inventory Score After 6 Months of Oral Contraceptive Use

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Bakircay University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes